CLINICAL TRIAL: NCT06697704
Title: Investigation of the Relationship Between Trunk Somatosensory Function, Trunk Control, and Thoracic Kyphosis in Children With Spastic Cerebral Palsy
Brief Title: Trunk Somatosensory Function, Trunk Control, and Thoracic Kyphosis in Children With Spastic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Gulce KALLEM SEYYAR, PhD, Assistant professor, Kutahya Health Sciences University
Other Study IDs: TYL-2023-127
Record Dates: First submitted 2024-03-15; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Spastic Cerebral Palsy
Keywords: cerebral palsy; trunk control; spinal curvature; somatosensory function
MeSH Terms: conditions — Cerebral Palsy; Spinal Curvatures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to investigate the relationship between trunk somatosensory function, trunk control, and thoracic kyphosis in children with cerebral palsy. The main questions it seeks to answer are:

* Is there a relationship between trunk somatosensory function and trunk control?
* Is there a relationship between trunk somatosensory function and thoracic kyphosis?
* Is there a relationship between trunk control and thoracic kyphosis?

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a heterogeneous disease group that occurs due to non-progressive lesion in the developing fetal or infant brain and causes constant and permanent impairments in movement, posture, and motor function. Sensory, perceptual, cognitive, communicative, and/or behavioral disorders, epilepsy, and secondary musculoskeletal problems may accompany motor disorders, the primary symptoms in CP. CP is one of the most common physical disabilities in childhood, with a reported prevalence of approximately 2.11 per 1,000 live births. Children with CP can be classified according to the type of motor impairment (physiological), the parts of the body affected (topographical), the etiology, the associated disorders, the neuroradiological findings (neuroanatomical), the therapy needs (therapeutic) and the functional abilities.The Surveillance of Cerebral Palsy in Europe (SCPE) classified CP as spastic, ataxic, and dyskinetic according to tone and dominant abnormal movement patterns. Spastic type is the most common form (70%).

Children with CP exhibit poor postural control due to abnormal muscle tone and movement patterns. This dysfunctional postural control causes limitations in gross motor skills such as balance and walking, upper extremity activities such as reaching, and oral-motor activities such as eating, swallowing, and speaking. Weak or inadequate postural control affects functional performance, participation in recreational and social activities, and society in children with CP.

The trunk is the reference point for postural control during stabilization and orientation. It is essential to ensure postural alignment, maintain postural balance, and interact with the environment (performing target-oriented activities). Trunk control refers to maintaining an upright posture, adjusting weight bearing, and performing selective movements while keeping the body's center of gravity within the support surface. In summary, trunk control is responsible for the stability and selective movements of the trunk. It is a precursor for ensuring optimal, targeted, selective, and dissociated movements of the head and extremities. Weak or inadequate trunk control is the basis of the limitations in the functional movements of children with CP. Although the pathophysiology is not progressive in CP, musculoskeletal disorders such as increased stiffness of spastic muscles, deterioration in spinal alignment, and joint contractures are observed with age. Weakness in trunk muscles in children and adults with CP may cause increased trunk extension and impaired spinal alignment in the sagittal plane in the sitting position. Impairment of spinal alignment negatively affects the motor function and activities of daily living of children with CP. It has also been found that the pathological alignment of the trunk and pelvis is associated with postural balance in children with CP.

Motor problems are often accompanied by sensory disorders in CP. Sensory disorders may also cause motor dysfunctions since sensory information for movement is impaired in children with CP. 90% of children with CP have sensory dysfunction. Recently, there has been an increasing interest in somatosensation among the senses in CP. The somatosensory system includes all peripheral and central components involved in the transmission and processing of sensory information from the superficial or cutaneous receptors and/or the musculoskeletal system and is closely related to the motor system. Somatosensory can be classified as tactile, proprioceptive, and pain sensation. It has been reported that somatosensory disorders are more common (97%) in children with unilateral CP.

Somatosensory deficits in CP have been associated primarily with damage to the developing brain and secondarily with motor disorders. Studies have also shown that motor impairments and somatosensory deficits are associated with children with CP. The literature shows that the relationship between somatosensory deficits and motor disorders in children with CP is primarily studied in the extremities (especially the upper extremities). A study evaluated trunk somatosensory function and motor impairments in children with CP. Only trunk proprioception (trunk position sense) was evaluated in this study among the somatosensations. A more comprehensive study, including tactile and pain sensations, has yet to be found. This study examines the relationship between trunk somatosensory function, trunk control, and thoracic kyphosis in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Received a diagnosis from a specialist doctor in the field
* Willing to participate, along with their family
* To be between the ages of 8-18
* The child with CP is able to tolerate the required test positions for the study

Exclusion Criteria:

* Received an additional diagnosis (down syndrome, autism, torticollis, etc.) other than CP from a specialist doctor in the field
* Has cognitive problems or attention disorders that prevent him/her from fulfilling the assessment instructions
* Botulinum Toxin A injection to the trunk or extremities, orthopedic surgery, and/or neurosurgery applications have been performed in the last six months.
* Having uncorrected visual and/or hearing problems

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with spastic cerebral palsy from city hospital and special education and rehabilitation center in Kocaeli and Sakarya, Turkey will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Light Touch, Tactile Sense | At baseline
  A measure of trunk somatosensory function, using a Semmes-Weinstein Monofilament (SWM) kit, consisting of 20 calibrated monofilaments in the prone position.
Two-Point Discrimination, Tactile Sense | At baseline
  A measure of trunk somatosensory function, using a discriminator in the prone position.
Vibration, Tactile Sense | At baseline
  A measure of trunk somatosensory function, using a 64 Hz tuning fork in the prone position.
Position Sense Reproduction, Proprioception Sense | At baseline
  A measure of trunk somatosensory function, using a digital inclinometer in a comfortable position with their hips and knees flexed to 90 degrees in the sitting position for the 30 degree trunk flexion and 10 degree trunk extension.
Pain Sense | At baseline
  A measure of trunk somatosensory function, using a dolorimeter for the pressure pain threshold in the prone position and the Visual Analogue Scale (VAS) for the pain severity.
Trunk Control | At baseline
  It was evaluated by the Trunk Control Measurement Scale (TCMS). TCMS is a reliable scale that assesses trunk control during functional activities, focusing on two components: static sitting balance and dynamic sitting balance. It consists of 15 items. Static sitting balance (items 1-5) evaluates trunk control while seated, while dynamic sitting balance includes selective movement control (items 6-12) for trunk movements in different planes, and dynamic reaching (items 13-15) for balance during reaching.The maximum scores are 20 for static sitting balance, 28 for selective movement control, and 10 for dynamic reaching. Higher scores indicate better trunk control performance.
Thoracic Kyphosis | At baseline
  Thoracic kyphosis in participants with cerebral palsy (CP) was assessed using a digital inclinometer. Participants sat comfortably on a Bobath bed with their hips and knees flexed at 90 degrees and feet on the floor. The T1 and T12 vertebrae were marked, and a dual digital inclinometer was attached to these points. The recorded value on the inclinometer's screen was noted in degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Gulce KALLEM SEYYAR, PT, PhD, Study Director — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brun C, Traverse E, Granger E, Mercier C. Somatosensory deficits and neural correlates in cerebral palsy: a scoping review. Dev Med Child Neurol. 2021 Dec;63(12):1382-1393. doi: 10.1111/dmcn.14963. Epub 2021 Jun 17. PMID 34145582
- [Background] Auld ML, Boyd RN, Moseley GL, Ware RS, Johnston LM. Impact of tactile dysfunction on upper-limb motor performance in children with unilateral cerebral palsy. Arch Phys Med Rehabil. 2012 Apr;93(4):696-702. doi: 10.1016/j.apmr.2011.10.025. Epub 2012 Feb 22. PMID 22360974
- [Background] McLean B, Taylor S, Valentine J, Carey L, Thornton A, Elliott C. Somatosensory discrimination impairment in children with hemiplegic cerebral palsy as measured by the sense_assess(c) kids. Aust Occup Ther J. 2021 Aug;68(4):317-326. doi: 10.1111/1440-1630.12729. Epub 2021 Mar 18. PMID 33738799
- [Background] Santana CAS, Dos Santos MM, de Campos AC. Interrelationships of Touch and Proprioception with Motor Impairments in Individuals with Cerebral Palsy: A Systematic Review. Percept Mot Skills. 2022 Jun;129(3):570-590. doi: 10.1177/00315125221093904. Epub 2022 Apr 22. PMID 35452588
- [Background] Monica S, Nayak A, Joshua AM, Mithra P, Amaravadi SK, Misri Z, Unnikrishnan B. Relationship between Trunk Position Sense and Trunk Control in Children with Spastic Cerebral Palsy: A Cross-Sectional Study. Rehabil Res Pract. 2021 Aug 19;2021:9758640. doi: 10.1155/2021/9758640. eCollection 2021. PMID 34462670